CLINICAL TRIAL: NCT00071747
Title: A Multi-Center, Double Blind, Placebo-controlled, Randomized, Parallel Group Evaluation of the Efficacy of a Flexible Dose of Lamotrigine Versus Placebo As Add-On Therapy In Schizophrenia
Brief Title: Clinical Study Of Schizophrenia in Both Men and Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCA30926
Record Dates: First submitted 2003-10-30; First posted 2003-10-31 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Schizophrenia
Keywords: schizophrenia; lamotrigine
MeSH Terms: conditions — Schizophrenia | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
The objective of this study is to evaluate the effectiveness of a marketed drug in the treatment of schizophrenia, as an add-on therapy to antipsychotics over a 12-week period. Subjects with schizophrenia who have been maintained on a stable dose of antipsychotics and who fulfill the screening entrance criteria will have an assessment 1-7 days after the first visit to confirm eligibility.

ELIGIBILITY:
Inclusion criteria:

* If female, must not be pregnant, or must be incapable of conceiving or be taking steps to prevent conception.
* Diagnosis of Schizophrenia
* Patients must be taking clozapine monotherapy or other atypical antipsychotic at least 3 months prior to this study.

Exclusion criteria:

* Patients who are currently taking or have taken antidepressant medication in the last month prior.
* Patients who are or have been suicidal or homicidal in the last 6 months.
* Patients with a history of autistic disorder or another pervasive developmental disorder
* Patients whose condition is due to the direct physiological effects of a substance (e.g. a drug of abuse, a medication) or a general medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176
Dates: Start 2003-08; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total score of the 7 items of the Positive and Negative Symptom Scale (PANSS) positive symptom subscale for lamotrigine vs. placebo at Week 12. | 12 Weeks

SECONDARY OUTCOMES:
Change from baseline in the PANSS total score at Week 12; Change from baseline in the Scale for the Assessment of Negative Symptoms (SANS) at Week 12; Change from baseline in the Clinical Global Impression-Severity of Illness (CGI-S) score at Week 12. | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (31):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Oceanside, California
  - GSK Investigational Site, Rosemead, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Maitland, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Granite City, Illinois
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Kenilworth, New Jersey
  - GSK Investigational Site, Orangeburg, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Butner, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Lyndhurst, Ohio
  - GSK Investigational Site, Norristown, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Bellaire, Texas
  - GSK Investigational Site, DeSoto, Texas
  - GSK Investigational Site, Midvale, Utah
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Goff DC, Keefe R, Citrome L, Davy K, Krystal JH, Large C, Thompson TR, Volavka J, Webster EL. Lamotrigine as add-on therapy in schizophrenia: results of 2 placebo-controlled trials. J Clin Psychopharmacol. 2007 Dec;27(6):582-9. doi: 10.1097/jcp.0b013e31815abf34. PMID 18004124
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: SCA30926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SCA30926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SCA30926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SCA30926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SCA30926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SCA30926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register